CLINICAL TRIAL: NCT06128057
Title: Comparing Trauma Associated Severe Hemorrhage "TASH" Score and Modified Traumatic Bleeding Severity Score "MTBSS" in Trauma Patients in Need for Massive Blood Transfusion in Assiut University Hospital
Brief Title: Comparing TASH Score and Modified TBSS in Trauma Patients in Need for Massive Blood Transfusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrhman Abouzeid, Resident, Assiut University
Other Study IDs: TASH score and MTBSS
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Massive Blood Transfusion in Trauma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood products — Massive blood transfusion

SUMMARY:
Evaluate And Compare predictive value of TASH Score And MTBBS In need for Massive Blood Transfusion

DETAILED DESCRIPTION:
Trauma is defined as a physical injury from an external source of sudden onset and severity, which require immediate medical attention.Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age group.

Approximately 5.8 million people die each year due to trauma related injuries, representing 8% of the worldwide mortality Polytrauma is a short verbal equivalent commonly used for severely injured patients usually with associated injury (i.e. two or more severe injuries in at least two different areas of the body), less often with a multiple injury (i.e. two or more severe injuries in one body area). Polytrauma patients usually have a much higher risk of mortalities and disabilities than the risk of expected mortalities in individual injuries patients.

Even though polytrauma can occur due to different causes such as road traffic accidents, fall from heights bullet injuries, suicide and homicide

.Yet the leading cause of traumatic related causes of death worldwide is road traffic accidents Egypt, in particular, has experienced an alarming increase in the burden of traumatic injuries. According to the World Health Organization In 2015 Egypt has one of the highest rates of road accidents worldwide, with more than 12,000 fatalities each year, one of the highest among Eastern Mediterranean countries. Although 90% of world's road trauma related fatalities occur in low- and middle-income countries, Injury

prevention and trauma care programs in these countries have remained deficient. The prediction of ongoing hemorrhage in severe trauma patients is challenging, and 14 scoring systems or algorithms have been developed to guide clinicians in this critical situation , the early identification of trauma patients with ongoing hemorrhage is pivotal for addressing their critical condition. Many of the scores are used in daily clinical practice and seem to be an interesting tool in the management of massive bleeding. The best scoring system would probably be one that combines superior accuracy in predicting the need for MT with an ease of use that would allow early identification of patients requiring Massive blood trasfusion.

Massive blood transfusion has often been defined as transfusion of ≥ 10 units of whole blood or red blood cells (RBC) within 24 h, as an approximation of the replacement of ≥ 1 total blood volume Or transfusion of ≥ 5 RBC units in 4 h, the replacement of ≥ 50% of total blood volume in 3 h, or ≥ 3 RBC units during any 1-h period in the first 24 h after hospital arrival The goal of this study is to reduce mortality by comparing between TASH and modified TBSS in prediction of need for massive blood transfusion in severe trauma patients .

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 years on both gender
* ISS ≥ 16

Exclusion Criteria:

* patients below 18 years
* patients with known bleeding disorders such as hemophilia or von Willebrand disease
* non trauma related bleeding : patients with severe hemorrhage unrelated to traumatic injury such as GI bleeding and ruptured aneurysm
* transfer from other facilities if their initial trauma records and scoring data are not available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-12-05 (Estimated); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Compare predictive value of TASH Score And MTBBS In need for Massive Blood Transfusion | Baseline
  Comparing odd number ( TASH score ) with even number (MTBSS ) in prediction for need for massive blood transfusion

REFERENCES:
- [Background] Ogura T, Lefor AK, Masuda M, Kushimoto S. Modified traumatic bleeding severity score: early determination of the need for massive transfusion. Am J Emerg Med. 2016 Jun;34(6):1097-101. doi: 10.1016/j.ajem.2016.02.072. Epub 2016 Mar 3. PMID 27021127
- [Background] Yucel N, Lefering R, Maegele M, Vorweg M, Tjardes T, Ruchholtz S, Neugebauer EA, Wappler F, Bouillon B, Rixen D; Polytrauma Study Group of the German Trauma Society. Trauma Associated Severe Hemorrhage (TASH)-Score: probability of mass transfusion as surrogate for life threatening hemorrhage after multiple trauma. J Trauma. 2006 Jun;60(6):1228-36; discussion 1236-7. doi: 10.1097/01.ta.0000220386.84012.bf. PMID 16766965
- [Background] Tonglet ML. Early Prediction of Ongoing Hemorrhage in Severe Trauma: Presentation of the Existing Scoring Systems. Arch Trauma Res. 2016 Jun 20;5(4):e33377. doi: 10.5812/atr.33377. eCollection 2016 Dec. PMID 28144603
- [Background] Bikbov B, Perico N, Remuzzi G. Mortality landscape in the global burden of diseases, injuries and risk factors study. Eur J Intern Med. 2014 Jan;25(1):1-5. doi: 10.1016/j.ejim.2013.09.002. Epub 2013 Sep 29. PMID 24084027
- [Background] Mitra B, Cameron PA, Gruen RL, Mori A, Fitzgerald M, Street A. The definition of massive transfusion in trauma: a critical variable in examining evidence for resuscitation. Eur J Emerg Med. 2011 Jun;18(3):137-42. doi: 10.1097/MEJ.0b013e328342310e. PMID 21164344
- [Background] Savage SA, Zarzaur BL, Croce MA, Fabian TC. Redefining massive transfusion when every second counts. J Trauma Acute Care Surg. 2013 Feb;74(2):396-400; discussion 400-2. doi: 10.1097/TA.0b013e31827a3639. PMID 23354230